CLINICAL TRIAL: NCT01532466
Title: The Effect of Priming Intravenous Rocuronium on Fentanyl-Induced Coughing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Huei-Chi Horng, MD, Principal Investigator, Taichung Armed Forces General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TC100-5
Record Dates: First submitted 2012-02-07; First posted 2012-02-14 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2011-12

CONDITIONS: Fentanyl-induced Coughing
Keywords: fentanyl-induced coughing, rocuronium
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocuronium, fentanyl-induced cough, normal saline (Experimental): All patients were given oxygen via a face mask. The patients were then administered with the following medications intravenously: the rocuronium group received rocuronium 0.06 mg kg-1 30 s before the injection of an IV fentanyl bolus (1.5 mcg kg-1, within 2 s).
  Interventions: Drug: Rocuronium
- Normal saline (No Intervention): All patients were given oxygen via a face mask. The patients were then administered with the following medications intravenously: the control group received the same volume of normal saline 30 s before the injection of an IV fentanyl bolus (1.5 mcg kg-1, within 2 s).

INTERVENTIONS:
Drug: Rocuronium — All patients were given oxygen via a face mask. The patients were then administered with the following medications intravenously: the rocuronium group received rocuronium 0.06 mg kg-1, and the control group received the same volume of normal saline 30 s before the injection of an IV fentanyl bolus (1.5 mcg kg-1, within 2 s).
  Arms: Rocuronium, fentanyl-induced cough, normal saline

SUMMARY:
An intravenous bolus of fentanyl often induces a cough reflex. This study investigates whether priming with rocuronium can attenuate fentanyl-induced coughing effectively.

DETAILED DESCRIPTION:
Fentanyl is widely used for analgesia and anesthesia because of its rapid onset, its intense analgesic effect, and is associated with lessened cardiovascular depression and low histamine release. Although the cough reflex is usually transient and self-limiting, it should be avoided in situations such as elevated intracranial, intraocular, or intra-abdominal pressure, and unstable hemodynamics.

The cause of FIC is unclear. One hypothesis is that vocal cord spasms might induce coughing because of fentanyl-induced muscle rigidity and histamine release. Muscle relaxants are commonly used to treat this condition. This study hypothesizes that priming muscle relaxants could prevent or suppress FIC. This study investigates whether the muscle relaxant rocuronium attenuates FIC effectively.

ELIGIBILITY:
Inclusion Criteria:

* 260 ASA I-II patients,
* aged between 18 and 80 years, and undergoing various elective surgeries at Taichung Armed Forces General Hospital.

Exclusion Criteria:

* a history of asthma,
* chronic cough,
* smoking,
* upper respiratory tract infection in the previous 2 weeks, and
* medication containing angiotensin-converting enzyme inhibitors or anesthetic premedication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of fentanyl-induced coughing | 2 minutes
  Following the fentanyl injection, another anesthetist who was blind to the pretreatment recorded the number of coughs for 1 min. The severity of coughing was graded as mild (1-2 times), moderate (3-5 times), or severe (> 5 times) based on the number of coughs within the 1 min following the fentanyl injection. Assisted mask ventilation with oxygen was supplied if desaturation occurred (SpO2 < 90%).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Shung Wong, PhD, Study Director — Cathay General Hospital
Locations (1):
- Taichung Armed Forces General Hospital, Taichung, Taiwan